CLINICAL TRIAL: NCT00622856
Title: The Cost-efficacy of Psychological Intervention for Strengthening Parental Authority Among Parents of Diabetic Adolescents With Poor Glycemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rmc004377ctil
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Diabetes
Keywords: diabetes; adolescents; psychological therapy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Psychosocial Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Psychological intervention for strengthening parental authority
  Interventions: Behavioral: psychological intervention
- 2 (Active Comparator): Diabetes education- 5 sessions with diabetes nurse, taking place once a week
  Interventions: Behavioral: Diabetes education
- 3 (No Intervention): Control group- regular treatment without any intervention

INTERVENTIONS:
Behavioral: psychological intervention — Psychological intervention
  Arms: 1
Behavioral: Diabetes education — 5 sessions with diabetes nurse
  Arms: 2

SUMMARY:
A three arms, open, randomized interventional study including 100 participants in order to evaluate the cost-efficacy of psychological intervention for strengthening parental authority among parents of diabetic adolescents with poor glycemic control.

All participants will be randomized into three groups:1.The first group will get a psychological treatment in order to strengthen the parent's authority. 2.The second group will get an education of a nurse and a dietician. 3.The third group will serve as a control group and will not go through an intervention.

The following data will be analyzed during the study: 1.Changes in HbA1c. 2.Changes in parents authority. 3.Changes in the diabetes treatment by the adolescents. 4.Consumption of health services. 5.The costs of all psychological treatments.

DETAILED DESCRIPTION:
A three arms, open, randomized interventional study including 100 participants in order to evaluate the cost-efficacy of psychological intervention for strengthening parental authority among parents of diabetic adolescents with poor glycemic control.

Objectives:

1. The primary purpose of the study is to evaluate the immediate effectiveness and the long run effectiveness of psychological intervention for strengthening parental authority among parents of diabetic adolescents with poor glycemic control.
2. To evaluate the cost as appose to the benefit of the psychological intervention.
3. To characterize the different variables in parent's attitude that improve their children's glycemic control.
4. To develop a therapy model for strengthening parent's authority which will be suitable for parents of diabetic adolescents.

Study design:

All participants in the study will be randomized to three different groups:

1. A treatment group that will go through psychological treatment to strengthen the parents authority.
2. A control group that will get an education of a nurse and a dietician
3. A control group that will not get any intervention. All groups will include parents of diabetic adolescents with poor glycemic control.

The following data will be analyzed during the study:

1. Changes in glycemic control will be measured by levels of HbA1C.
2. Changes in the diabetes treatment by the adolescents will be measured by adherence to insulin injections, the number of times a day in which the patient checked his blood glucose values, number of visits in the clinic and psychological questionnaires.
3. Consumption of health services
4. Changes in parents attitude and changes in the wellbeing of the diabetic adolescents and their parents will be based on questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Parents of adolescents between the ages of 10-18
2. More than one year diabetes
3. Adolescent's HbA1c>8

Exclusion Criteria:

1. Adolescents or parents of adolescents that are mentally retarded.
2. Another chronic disease besides diabetes.
3. Adolescents that are taking medications that might disturb their glycemic control.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
HbA1c | Every three months
adherence to treatment | before the intervention, after the intervention and at the end of the study
consumption of health services | during the study and at the end of the study

SECONDARY OUTCOMES:
Changes in the wellbeing of adolescents and their parents | In the beginning of the study, at the end of the intervention and after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Meyerovitch, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Schneider Children's Medical Center, Petah Tikva, Israel

REFERENCES:
- [Derived] Yackobovitch-Gavan M, Meshy-Tamir R, Nagelberg N, Phillip M, Meyerovitch J. Psychosocial factors associated with depressive mood in Israeli obese adolescents. J Health Psychol. 2014 Apr;19(4):574-84. doi: 10.1177/1359105313475901. Epub 2013 Mar 11. PMID 23479303